CLINICAL TRIAL: NCT00168103
Title: Human Pasteurized C1 Esterase Inhibitor Concentrate (CE1145) in Subjects With Congenital C1-INH Deficiency and Acute Abdominal or Facial HAE Attacks
Brief Title: Human C1 Esterase Inhibitor (C1-INH) in Subjects With Acute Abdominal or Facial Hereditary Angioedema (HAE) Attacks
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Global Head Clinical Research & Development, CSL Behring
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CE1145_3001; 2004-001186-17 (EudraCT Number)
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Results first posted 2010-08-24 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2011-02

CONDITIONS: Hereditary Angioedema
Keywords: C1 Inhibitor; Hereditary angioedema; Acute HAE attack
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — Complement C1 Inhibitor Protein

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- C1-INH 10 U/kg bw (Experimental): 10 Units (U)/kg body weight (bw) dose
  Interventions: Biological: C1 Esterase Inhibitor
- C1-INH 20 U/kg bw (Experimental): 20 U/kg bw dose
  Interventions: Biological: C1 Esterase Inhibitor
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: C1 Esterase Inhibitor — Single application of C1-INH administered intravenously by slow injection or infusion at a recommended rate of 4mL/min.
  Other Names: Berinert; Berinert P; CE1145
  Arms: C1-INH 10 U/kg bw; C1-INH 20 U/kg bw
Biological: Placebo — Single application of physiological saline solution equivalent to the volume calculated for subjects in the C1-INH 20 U/kg bw arm.
  Other Names: Physiological saline solution
  Arms: Placebo

SUMMARY:
HAE is a rare disorder characterized by functional C1 esterase inhibitor deficiency. If not treated adequately, the acute attacks of HAE can be life-threatening and may even result in fatalities, especially in case of swelling of the larynx. This clinical Phase 2/Phase 3 study was designed to provide clinically relevant data on dosing, efficacy and safety in subjects with HAE.

DETAILED DESCRIPTION:
For each subject, only a single abdominal or facial attack was treated and evaluated. After receiving treatment, subjects were observed for a minimum of 4 hours, after which they could be discharged from the study center if they reported onset of symptom relief. Starting from 4 hours after treatment, subjects who reported insufficient or no symptom relief could receive a second dose of double-blind treatment (called "rescue medication") as follows: C1-INH 20 U/kg bw for subjects initially receiving placebo, C1-INH 10 U/kg bw for subjects initially receiving C1-INH 10 U/kg bw, and placebo for subjects initially receiving C1-INH 20 U/kg bw.

The study was defined to be successful if the primary outcome measure and at least one of the secondary outcome measures were met in the comparison between the C1-INH 20 U/kg bw group and the Placebo group.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented congenital C1-INH deficiency
* Acute facial or abdominal HAE attack

Key Exclusion Criteria:

* Acquired angioedema
* Treatment with any other investigational drug within the last 30 days before study entry
* Treatment with any C1-INH concentrate within the previous 7 days

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2005-06; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Clinical R&D, Study Director — CSL Behring
Locations (36):
- United States (17):
  - Study Site, Granada Hills, California
  - Study Site, Weston, Florida
  - Study Site, Atlanta, Georgia
  - Study Site, Idaho Falls, Idaho
  - Study Site, Chicago, Illinois
  - Study Site, Shreveport, Louisiana
  - Study Site, Boston, Massachusetts
  - Study Site, Plymouth, Minnesota
  - Study Site, Omaha, Nebraska
  - Study Site, The Bronx, New York
  - Study Site, Cincinnati, Ohio
  - Study Site, Tulsa, Oklahoma
  - Study Site, Eugene, Oregon
  - Study Site, Hershey, Pennsylvania
  - Study Site, Rapid City, South Dakota
  - Study Site, Dallas, Texas
  - Study Site, Bellingham, Washington
- Study Site, Buenos Aires, Argentina
- Study Site, Westmead, Australia
- Bulgaria (2):
  - Study Site, Plovdiv
  - Study Site, Sofia
- Canada (2):
  - Study Site, Edmonton
  - Study Site, Ottawa
- Study Site, Brno, Czechia
- Study Site, Budapest, Hungary
- Study Site, Tel Litwinsky, Israel
- Study Site, Skopje, North Macedonia
- Poland (2):
  - Study Site, Grodzisk Mazowiecki
  - Study Site, Krakow
- Study Site, Târgu Mureş, Romania
- Russia (3):
  - Study Site 1, Moscow
  - Study Site 2, Moscow
  - Study Site 3, Moscow
- Study Site, Madrid, Spain
- Study Site, Gothenburg, Sweden
- Study Site, London, United Kingdom

REFERENCES:
- [Background] Bernstein JA, Ritchie B, Levy RJ, Wasserman RL, Bewtra AK, Hurewitz DS, Obtulowicz K, Reshef A, Moldovan D, Shirov T, Grivcheva-Panovska V, Kiessling PC, Keinecke HO, Craig TJ. Hereditary angioedema: Validation of the end point time to onset of relief by correlation with symptom intensity. Allergy Asthma Proc. 2011 Jan-Feb;32(1):36-42. doi: 10.2500/aap.2011.32.3404. PMID 21262096
- [Result] Craig TJ, Levy RJ, Wasserman RL, Bewtra AK, Hurewitz D, Obtulowicz K, Reshef A, Ritchie B, Moldovan D, Shirov T, Grivcheva-Panovska V, Kiessling PC, Keinecke HO, Bernstein JA. Efficacy of human C1 esterase inhibitor concentrate compared with placebo in acute hereditary angioedema attacks. J Allergy Clin Immunol. 2009 Oct;124(4):801-8. doi: 10.1016/j.jaci.2009.07.017. Epub 2009 Sep 19. PMID 19767078
- [Derived] Craig TJ, Rojavin MA, Machnig T, Keinecke HO, Bernstein JA. Effect of time to treatment on response to C1 esterase inhibitor concentrate for hereditary angioedema attacks. Ann Allergy Asthma Immunol. 2013 Sep;111(3):211-5. doi: 10.1016/j.anai.2013.06.021. Epub 2013 Jul 16. PMID 23987198
- [Derived] Bernstein JA, Ritchie B, Levy RJ, Wasserman RL, Bewtra AK, Hurewitz DS, Obtulowicz K, Reshef A, Moldovan D, Shirov T, Grivcheva-Panovska V, Kiessling PC, Schindel F, Craig TJ. Population pharmacokinetics of plasma-derived C1 esterase inhibitor concentrate used to treat acute hereditary angioedema attacks. Ann Allergy Asthma Immunol. 2010 Aug;105(2):149-54. doi: 10.1016/j.anai.2010.06.005. PMID 20674826

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multinational study enrolling subjects at 36 study centers in 15 countries.
Pre-assignment Details: A screening visit was performed before the subject presented with an hereditary angioedema (HAE) attack at the study center. Study entry was defined to occur with administration of study treatment.
  One subject enrolled received study treatment without being randomized and is listed separately in the participant flow.
Groups:
- C1-INH 10 U/kg bw: Includes all subjects enrolled and randomized to the C1 Esterase Inhibitor (C1-INH) 10 Units (U)/kg body weight (bw) arm.
- C1-INH 20 U/kg bw: Includes all subjects enrolled and randomized to the C1-INH 20 U/kg bw arm.
- Placebo: Includes all subjects enrolled and randomized to the Placebo arm.
- Not Randomized: Includes one subject enrolled who was not randomized but received treatment with 20 U/kg bw C1-INH.
Period: Overall Study
Arm/Group | C1-INH 10 U/kg bw | C1-INH 20 U/kg bw | Placebo | Not Randomized
Started | 40 | 43 | 42 | 1
Completed | 38 (1 randomized subject received open-label rescue medication before receiving randomized treatment.) | 38 | 41 | 1
Not Completed | 2 | 5 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- C1-INH 10 U/kg bw: Baseline characteristics were calculated only for the intention to treat (ITT) and per protocol (PP) analysis populations, not for all enrolled subjects. Baseline data presented here are for subjects included in the ITT population. One (1) subject enrolled and randomized to the C1-INH 10 U/kg bw group was excluded from the ITT analysis population.
- C1-INH 20 U/kg bw: Baseline data presented here are for subjects included in the ITT population. All subjects enrolled and randomized to the C1-INH 20 U/kg bw arm were included in the ITT analysis population.
- Placebo: Baseline data presented here are for subjects included in the ITT population. All subjects enrolled and randomized to the Placebo arm were included in the ITT analysis population.
- Total: Total of all reporting groups
Arm/Group | C1-INH 10 U/kg bw | C1-INH 20 U/kg bw | Placebo | Total
Number analyzed (Participants) | 39 | 43 | 42 | 124
Age, Customized [Number; unit: participants]
  3 to < 12 years | 0 | 1 | 2 | 3
  12 to < 17 years | 3 | 4 | 3 | 10
  17 to < 65 years | 35 | 35 | 37 | 107
  >= 65 years | 1 | 3 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.1 (12.77) | 34.6 (14.91) | 31.5 (13.57) | 33.1 (13.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 30 | 28 | 84
  Male | 13 | 13 | 14 | 40
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 36 | 38 | 37 | 111
  Black | 0 | 3 | 1 | 4
  Hispanic | 2 | 2 | 1 | 5
  Asian | 1 | 0 | 2 | 3
  American Indian or Alaskan Native | 0 | 0 | 1 | 1
Intensity of Baseline HAE Attack [Number; unit: Participants]
  Moderate | 32 | 27 | 26 | 85
  Severe | 7 | 16 | 16 | 39
Primary Disease Characteristic [Number; unit: Participants] — Type I HAE (common form genotype): An impaired synthesis and an elevated turnover of a normal and functionally active C1-INH molecule occurs, causing a reduction in the availability of functionally active C1-INH to levels of 5% to 30% of normal.
  Type II HAE (variant form genotype): Normal levels of a functionally impaired C1-INH molecule are synthesized while the normal form of C1-INH is considerably reduced in the circulation.
  Participants
    Type I HAE | 35 | 35 | 38 | 108
    Type II HAE | 3 | 8 | 4 | 15
    Missing | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Time to Start of Relief of Symptoms From HAE Attack
Description: The start of symptom relief was determined by subject self-assessment. Time to start of symptom relief was set to 24 hours if the subject received rescue medication (blinded study medication, narcotic analgesics, antiemetics, open-label C1-INH, or fresh frozen plasma) at any time point after the start of study treatment but before start of relief.
Time Frame: Up to 24 h after start of study treatment
Population: Analysis was based on the ITT population which included all subjects receiving any portion of the randomized study medication.
Measure: Median (Full Range); unit: Hours
Groups:
- C1-INH 10 U/kg bw: Includes all subjects enrolled and randomized to the C1-INH 10 U/kg bw arm.
Arm/Group | C1-INH 10 U/kg bw | C1-INH 20 U/kg bw | Placebo
Number analyzed (Participants) | 39 | 43 | 42
Hours | 1.17 (10.513) [0.17 to 24.00] | 0.5 (8.202) [0.17 to 24.00] | 1.5 (11.481) [0.20 to 24.00]
Statistical Analysis 1: Comparison: C1-INH 20 U/kg bw vs Placebo; Test type: Superiority or Other; p = 0.0025, Wilcoxon (Mann-Whitney) — 1-sided P-value. The a priori threshold was 0.024 (overall Type 1 error 0.025 adjusted for alpha spending for an interim analysis); 1-sided; Median Difference (Final Values) = -0.525, 95% CI 2-sided [-2.217 to -0.033] — The median difference was estimated by the Hodges-Lehmann estimate

2. Secondary Outcome: Number of Subjects With Worsened Intensity of Clinical HAE Symptoms
Description: Includes any worsening of intensity of at least 1 of the HAE symptoms present at baseline. Routinely checked symptoms included pain, nausea, vomiting, cramps, and diarrhea.
Time Frame: Baseline and between 2 and 4 h after start of study treatment
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | C1-INH 10 U/kg bw | C1-INH 20 U/kg bw | Placebo
Number analyzed (Participants) | 39 | 43 | 42
Subjects | 8 | 2 | 13
Statistical Analysis 1: Comparison: C1-INH 20 U/kg bw vs Placebo; Worsened intensity was evaluated between 2 and 4 hours after start of study treatment relative to baseline for at least 1 of the HAE symptoms present at baseline; Test type: Superiority or Other; p = 0.0014, Fisher Exact — 1-sided P-value. The a priori threshold for significance was 0.1 (trend); 1-sided; Odds Ratio (OR) = 0.1088, 80% CI 2-sided [0.0392 to 0.3023] — The Odds Ratio was calculated as C1-INH 20 U/kg bw (numerator) versus Placebo (denominator)

3. Other Pre Specified Outcome: Time to Complete Resolution of All HAE Symptoms, Including Pain
Description: Complete resolution of symptoms was determined by subject self-assessment.
Time Frame: Up to 24 h after start of study treatment
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | C1-INH 10 U/kg bw | C1-INH 20 U/kg bw | Placebo
Number analyzed (Participants) | 39 | 43 | 42
Hours | 20.00 (494.230) [0.47 to 1486.17] | 4.92 (314.347) [0.47 to 1486.17] | 7.79 (382.815) [0.33 to 1486.17]
Statistical Analysis 1: Comparison: C1-INH 20 U/kg bw vs Placebo; This was an exploratory analysis; Test type: Superiority or Other; p = 0.0237, Wilcoxon (Mann-Whitney) — 1-sided, exploratory test; 1-sided; Median Difference (Final Values) = -3.292, 80% CI 2-sided [-5.150 to -1.050] — The median difference was estimated by the Hodge-Lehmann estimate

4. Other Pre Specified Outcome: Number of Subjects Receiving Rescue Study Medication
Time Frame: Within 4 h after start of study treatment
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | C1-INH 10 U/kg bw | C1-INH 20 U/kg bw | Placebo
Number analyzed (Participants) | 39 | 43 | 42
Subjects | 13 | 8 | 24
Statistical Analysis 1: Comparison: C1-INH 20 U/kg bw vs Placebo; This was an exploratory analysis; Test type: Superiority or Other; Odds Ratio (OR) = 0.1714, 95% CI 2-sided [0.0642 to 0.4575] — The Odds Ratio was calculated as C1-INH 20 U/kg bw (numerator) versus Placebo (denominator)

5. Secondary Outcome: Number of Vomiting Episodes
Time Frame: Within 4 h after start of study treatment
Population: as for outcome 1
Measure: Median (Full Range); unit: Episodes per subject
Arm/Group | C1-INH 10 U/kg bw | C1-INH 20 U/kg bw | Placebo
Number analyzed (Participants) | 39 | 43 | 42
Episodes per subject | 0 (0.77) [0 to 4] | 0 (0.41) [0 to 2] | 0 (2.59) [0 to 16]
Statistical Analysis 1: Comparison: C1-INH 20 U/kg bw vs Placebo; Test type: Superiority or Other; p = 0.0329, Wilcoxon (Mann-Whitney) — 1-sided P-value. The a priori threshold for significance was 0.1 (trend); 1-sided

ADVERSE EVENTS:
Time Frame: AEs for each study arm are reported for the first 4 hours after start of study treatment.
Description: Safety data were analyzed according to the actual treatment received. The analysis of AEs within 4 hours of the start of initial treatment permits an unbiased comparison of treatment groups without the confounding effect of any rescue medication.
Groups:
- C1-INH 10 U/kg bw: Includes subjects receiving 10 U/kg bw C1-INH and no rescue study medication within 4 hours after the start of the initial treatment.
- C1-INH 20 U/kg bw: Includes subjects receiving 20 U/kg bw C1-INH and no rescue study medication within 4 hours after the start of the initial treatment (n=43). An additional 3 subjects not randomized to but treated with 20 U/kg bw C1-INH in this time period were also included in this group for the safety analysis.
- Placebo: Includes subjects receiving Placebo and no rescue study medication within 4 hours after the start of the initial treatment.
Arm/Group | C1-INH 10 U/kg bw | C1-INH 20 U/kg bw | Placebo
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/46 | 0/41
Other Adverse Events (participants affected / at risk) | 10/39 | 10/46 | 18/41
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | C1-INH 10 U/kg bw (N=39) | C1-INH 20 U/kg bw (N=46) | Placebo (N=41)
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 4
Dysgeusia (Nervous system disorders) | 1 | 2 | 0
Edema peripheral (General disorders) | 1 | 1 | 0
Face edema (General disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 2
Lip swelling (Gastrointestinal disorders) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 3 | 5
Pain (General disorders) | 4 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 3

LIMITATIONS AND CAVEATS:
A test for futility of the C1-INH 10 U/kg bw group conducted during a planned interim analysis led to ceasing recruitment for the C1-INH 10 U/kg bw group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must provide a copy of any results communication to the sponsor for review at least 30 days prior to public release. The sponsor may request any changes necessary to prevent forfeiture of patent rights to data not in the public domain. For a multi-center study, the investigator must wait (i) at least 1 year after the study is completed at all sites or (ii) until notified by the sponsor that no multi-center publication is planned before seeking publication review.